CLINICAL TRIAL: NCT02914249
Title: Low-calorie Diet Combined With Orange Juice Results in Weight Loss: Randomized Controlled Trial
Brief Title: Effect of Low-calorie Diet and Orange Juice on Body Weight and Metabolic Parameters of Obese Subjects
Acronym: LCD-OJ-OBESE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Collaborators: National Association of Exporters of Citrus Juices (Other); Citrosuco Company (Industry)
Responsible Party: Principal Investigator, Thais Cesar, Principal Investigator, São Paulo State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SaoPSU1
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
Keywords: Orange juice; Low-calorie diet; Body composition; Weight-loss; Metabolic biomarkers; Obese
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orange juice (Experimental): Orange juice: thirty-nine obese individuals were submitted to a low-caloric diet (500 kcal/d of energy restriction) plus 100% orange juice (500 mL/d) during 12 weeks.
  Interventions: Other: Orange juice (500 mL/d)
- Control (No Intervention): Control: thirty-nine obese individuals were submitted to a low-caloric diet (500 kcal/d of energy restriction) during 12 weeks.

INTERVENTIONS:
Other: Orange juice (500 mL/d) — Nutritionists prescribed a low-calorie diet that was estimated from total energy expenditure (TEE) for each individual minus 500 kcal per day (30% TEE). Both groups had the same diet plan based on individual weight. The dietary plan was composed of six meals/day: breakfast (fat-free milk and coffee; whole-grain bread with margarine, and an apple); snack 1 (250 mL OJ / banana and free-fat yogurt); lunch (brown rice, beans, grilled lean meat, salad, cooked vegetables); snack 2 (250 mL OJ / free-fat yogurt with oatmeal); dinner (brown rice, beans, grilled lean meat, cooked vegetables and salad); and snack 3 (salty crackers or oat cookies, tea without sugar). Body composition measurements were collected (monthly); blood samples and dietary questionnaires (every two weeks).
  Arms: Orange juice

SUMMARY:
This study aimed to verify if combination of a low calorie diet and orange juice consumption results in weight loss and ameliorates metabolic obesity-related biomarkers.

DETAILED DESCRIPTION:
Seventy-eight obese subjects aged 36 ± 1 years and BMI of 33 ± 3 kg were randomly divided into two parallel groups: (1) orange juice (n = 39), composed of individuals subjected to a diet low caloric diet and plus intake of 500 ml orange juice; (2) control (n = 39) composed of individuals subjected to a diet low in calories. The recruitment process began in September 2015, the intervention was carried out from October 2015 to January 2016, and the data analysis started in February 2016. The sample number took into account variances on body weight with a type I error α = 0.05 and a type II error β = 0.2 (80% power). The minimum sample size should have 36 individuals per group (n = 72), considering an approximately 15% dropout rate. Thus, the final sample size of study was constituted by 39 individuals per group (n = 78). Primary and secondary endpoints were the reduction of weight and modification of the levels of obesity-related metabolic biomarkers, respectively. Normality and homogeneity of data were tested. T-test was conducted to identify possible differences between OJ and control groups at baseline. A linear mixed-effects model was apply to determine the time effect within and between groups (post hoc), and P significance was set up ≤ 0.05. The assessment of body composition, metabolic biomarkers and food intake were analyzed over a 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* 30 > BMI < 40 kg/m2

Exclusion Criteria:

* Dieting last year,
* Use of drugs, vitamins and dietary supplements
* Alcohol consumption (> 20 g alcohol/d)
* Intense physical activity (> 5 hours/week).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Body-weight | 12 weeks

SECONDARY OUTCOMES:
Body mass index (BMI) | 12 weeks
Body lean mass | 12 weeks
Body fat mass | 12 weeks
Percentage of body fat | 12 weeks
Ratio waist/hip | 12 weeks
Glucose | 12 weeks
Insulin | 12 weeks
Homeostatic Model assessment of Insulin Resistance | 12 weeks
Total cholesterol | 12 weeks
LDL-cholesterol | 12 weeks
HDL-cholesterol | 12 weeks
Non-HDL-cholesterol | 12 weeks
Triglycerides | 12 weeks
hsCRP | 12 weeks
Alkaline phosphatase | 12 weeks
Aspartate transaminase | 12 weeks
Alanine transaminase | 12 weeks
Gamma-glutamyl transferase | 12 weeks
Antioxidant capacity (ABTS) | 12 weeks
Lipid peroxidation (TBARS) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thais B Cesar, Ph.D., Principal Investigator — Sao Paulo State University "Julio de Mesquita Filho" (UNESP)